CLINICAL TRIAL: NCT06897410
Title: Reforça't: A Randomized Community Clinical Trial With a Social and Healthcare Approach to Improve Functional Outcomes in Patients With Chronic Cardiac, Respiratory, or Mixed Conditions After Hospital Discharge
Brief Title: Reforça't: A Community, Social, and Healthcare Program for Patients With Cardiorespiratory Conditions Upon Hospital Discharge
Acronym: R't
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corporació de Salut del Maresme i la Selva (Other)
Collaborators: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Griselda Manzano Monfort, Head of Hospital At Home Unit at Corporació de Salut del Maresme i la Selva (CSMS). Postdoctoral researcher at Digital Health Research Group (IDIBGI-CSMS), Corporació de Salut del Maresme i la Selva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R't
Record Dates: First submitted 2025-03-06; First posted 2025-03-26 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Chronic Obstructive Lung Disease (COLD); Heart Failure
Keywords: Patient Readmission; COLD; Heart Failure; Frail elderly; Multidisciplinary care team
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure | interventions — Aging

STUDY DESIGN:
Intervention Model Description: Randomized Intervention Study, control vs intervention group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): Standard Follow-up under hospital at home regime in our institution
- Intervention Group (Experimental): Presential Follow-up by a multidisciplinary team
  Interventions: Other: Interdisciplinary Program for Post-Hospitalization / Hospital at home Management and Long-Term Outcomes in Older Adults with Chronic Cardiorespiratory Condition

INTERVENTIONS:
Other: Interdisciplinary Program for Post-Hospitalization / Hospital at home Management and Long-Term Outcomes in Older Adults with Chronic Cardiorespiratory Condition — Intervention Phase 1: Feasibility Assessment Duration: January 7, 2025 - January 11, 2025 Participants: 10-15 patients
  Description:
  All involved services will be available to address and resolve potential issues.
  The objective is to assess the feasibility of the program, ensuring that the intervention can be implemented as planned and identifying any practical or logistical challenges.
  Phases 2 & 3: Comprehensive Intervention Duration: January 12, 2025 - June 30, 2025 Participants: 200 patients
  Description:
  Full-scale implementation of the intervention. Includes interdisciplinary care, home follow-ups, therapeutic optimization, functional rehabilitation, health education, and psychosocial support.
  Phase 4: Long-Term Follow-Up Duration: April 7, 2025 - June 30, 2026 Participants: 200 patients
  Description:
  Follow-up assessments at 3, 6, 9, and 12 months post-intervention. Evaluates hospital readmissi
  Arms: Intervention Group

SUMMARY:
The goal of this randomized clinical trial is to determine whether an interdisciplinary, community-based intervention can reduce 30-day hospital readmissions and improve functional outcomes in patients aged 65 or older with chronic cardiac, respiratory, or mixed conditions following hospital discharge.

The main questions it aims to answer are:

Can the Reforça't program reduce 30-day hospital readmission rates to 25% compared to standard care? Does participation in Reforça't improve functional outcomes, medication adherence, quality of life, and mortality rates in this patient population?

Researchers will compare patients enrolled in Reforça't (intervention group) with those receiving standard care (control group) to determine whether the program leads to lower readmission rates, improved health outcomes, and higher cost-effectiveness.

Participants will:

Undergo a pre- and post-intervention assessment (30 days post-discharge). Receive comprehensive, interdisciplinary care integrating medical, social, and rehabilitation services.

Be monitored for 12 months to assess readmissions, survival, nursing home admissions, and overall well-being.

ELIGIBILITY:
Inclusion Criteria:

* Users admitted to the Polivalent Observation Units, Internal Medicine, or Hospital at home.
* Individuals aged 65 years or older.
* Hospital admission due to decompensation of a cardiac, respiratory, or mixed condition.
* Place of residence within the health coverage area of Sant Jaume de Calella Hospital - Corporació de Salut del Maresme i la Selva.
* Willingness to participate in the study as gathered by the signing of an informed consent document

Exclusion Criteria:

* Users institutionalized in a nursing home
* Users already enrolled in home care programs
* Users in the Advanced Chronic Care Model program with a limited life prognosis
* Users on the waiting list for organ transplantation
* Users with language barriers
* Users with a GDS (Global Deterioration Scale) score of 5 or higher
* Users who have already been included in the Reforça't program

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Reduction of the Readmission Rate in the Intervention Group | 30 days after hospital discharge
  The investigators aim for the intervention to result in a 20% reduction of the readmission rate among users included in the experimental group
Reduction of mortality, readmission and nursing home admission | 3, 6, 9, and 12 months after hospital discharge

SECONDARY OUTCOMES:
Reduction in Frailty Index Score | 30 days after hospital discharge
Reduction of the mortality rate | 30 days after hospital discharge
Reduction in the number of inappropriate prescriptions | 30 days after hospital discharge
Increase in pharmacotherapeutic adherence | 30 days after hospital discharge
  The investigators will conduct the spanish version of the Adherence to Refills and Medications Scale (ARMS-e).
  Per this scale, high scores indicate low therapeutic adherence. Subjects are classified into high adherence (scores from 0 to 16), intermediate adherence (scores from 17 to 32), and low adherence (scores from 33 to 48).
  - Expected experimental range values: 12 - 48
Reduction in functional deterioration | 30 days after hospital discharge
  The investigators will measure Barthel and Lawton scores to determine functional activity.
  Barthel index indicates the ability to perform daily tasks autonomously. Higher Barthel index equals higher degree of autonomy. Values range from 0 to 100. Scores lower than 20 indicate total dependence, between 20 and 35 equal severe dependence, between 50 and 55 indicate moderate dependence, between 60 and 90 indicate light dependent, and higher than 95 indicate autonomy.
  Lawton and Brody scores measure the degree of autonomy in the performance of instrumental activities of daily living. Values range from 0 to 8, with higher score indicating higher autonomy.
Reduction in the risk of falls | 30 days after hospital discharge
  The investigators will assess the Downton score. This measure is expected to decrease in the intervention group. Values range from 0 to 11, where higher score equals higher risk. Starting at 3, the values are considered to indicate relevant risk of fall.
Increase in physical function | 30 days after hospital discharge
  The investigators will conduct Short Physical Performance Battery (SPPB) and assess Daniels score, to determine subjects' physical function.
  * SPPB values range from 0 to 12. Higher score equals higher physical function (less frailty). Values lower than 10 indicate clinically relevant frailty and risk of falls
  * Daniel's score values range from 0 to 5. Higher values indicate higher strength for the evaluated muscle. Each value indicates; i) 0-absence of contraction, ii) 1- contraction without movement, iii) 2- movement with gravity eliminated iv) 3-full range of motion against gravity, v) 4-full range of motion against moderate resistance, vi) 5-full range of motion against maximum resistance
Increase in the number of beneficiaries of social prescribing or community referrals | 30 days after hospital discharge
Obtain positive patient satisfaction | 30 days after hospital discharge
  The investigators will administer ad hoc patient satisfaction surveys. Results will be numerical, from 0 (min) to 10 (max). Average above 7 will be considered a success, although results greater than 5 will be deemed satisfactory.
Reduction or delay in institutionalization in nursing homes among users | 30 days after hospital discharge
Reduction in Zarit Score for caregiver burden | 30 days after hospital discharge
  The investigators will conduct Zarit Burden Interviews (ZBI) on caregivers for patients included in the study. Specifically, the short ZBI-7 will be assessed. It consists of 7 items, each item scoring from 1 to 5. Per this score, the higher the score equals a higher caregiver burden. Thus, a reduction in the Zarit Score for caregivers included in the study is expected.
  The obtained values per caregiver range from 7 to 35, and a total score of 17 or higher is considered excessive burden.
Reduction in the risk of social isolation | 30 days after hospital discharge
  The investigators will determine OSSS-3 score for patients included in the study.
  Higher scores determine higher perception of social support. Scores between 3 and 8 equal low social support, between 9 and 11 intermediate social support, and higher scores equal high social support. The patients included in the study are expected to range between 3 and 14.
Increase in emotional well-being | 30 days after hospital discharge
  The investigators will conduct the short Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) to measure subject emotional well-being. Higher scores indicate better emotional wellbeing. A score lower than 26 is considered to relate to emotional discomfort. The patients included are expected to range between 7 and 35 in score (35 is the maximum score for this short version).
Increase in the smoking cessation rate | 30 days after hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Comarcal de Calella - Corporació de Salut del Maresme i la Selva, Calella, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aranda-Gallardo M, Morales-Asencio JM, Canca-Sanchez JC, Morales-Fernandez A, Enriquez de Luna-Rodriguez M, Moya-Suarez AB, Mora-Banderas AM, Perez-Jimenez C, Barrero-Sojo S. [Consequences of errors in the translation of questionnaires: Spanish version of Downton index]. Rev Calid Asist. 2015 Jul-Aug;30(4):195-202. doi: 10.1016/j.cali.2015.04.003. Epub 2015 Jun 9. Spanish. PMID 26068277
- [Background] Castellvi P, Forero CG, Codony M, Vilagut G, Brugulat P, Medina A, Gabilondo A, Mompart A, Colom J, Tresserras R, Ferrer M, Stewart-Brown S, Alonso J. The Spanish version of the Warwick-Edinburgh mental well-being scale (WEMWBS) is valid for use in the general population. Qual Life Res. 2014 Apr;23(3):857-68. doi: 10.1007/s11136-013-0513-7. Epub 2013 Sep 5. PMID 24005886
- [Background] Kocalevent RD, Berg L, Beutel ME, Hinz A, Zenger M, Harter M, Nater U, Brahler E. Social support in the general population: standardization of the Oslo social support scale (OSSS-3). BMC Psychol. 2018 Jul 17;6(1):31. doi: 10.1186/s40359-018-0249-9. PMID 30016997
- [Background] Zamora-Sanchez JJ, Zabaleta-Del-Olmo E, Gea-Caballero V, Julian-Rochina I, Perez-Tortajada G, Amblas-Novellas J. [Convergent and discriminative validity of the Frail-VIG index with the Braden scale in people cared for in home care]. Rev Esp Geriatr Gerontol. 2022 Mar-Apr;57(2):71-78. doi: 10.1016/j.regg.2021.12.003. Epub 2022 Mar 17. Spanish. PMID 35307198
- [Background] Charlson ME, Charlson RE, Peterson JC, Marinopoulos SS, Briggs WM, Hollenberg JP. The Charlson comorbidity index is adapted to predict costs of chronic disease in primary care patients. J Clin Epidemiol. 2008 Dec;61(12):1234-1240. doi: 10.1016/j.jclinepi.2008.01.006. Epub 2008 Jul 10. PMID 18619805
- [Background] Pinzon-Pulido S, Garrido Pena F, Reyes Alcazar V, Lima-Rodriguez JS, Raposo Triano MF, Martinez Domene M, Alonso Trujillo F. [Predictors of institutionalization of elderly persons in dependency situation in Andalusia]. Enferm Clin. 2016 Jan-Feb;26(1):23-30. doi: 10.1016/j.enfcli.2015.08.003. Epub 2015 Sep 9. Spanish. PMID 26363992
- [Background] Acosta-Benito MA, Martin-Lesende I. [Frailty in primary care: Diagnosis and multidisciplinary management]. Aten Primaria. 2022 Sep;54(9):102395. doi: 10.1016/j.aprim.2022.102395. Epub 2022 Jun 11. Spanish. PMID 35700618
- [Background] Bayona Huguet X, Limon Ramirez E, Cegri Lombardo F. [Proposals for home care of the XXI century]. Aten Primaria. 2018 May;50(5):264-266. doi: 10.1016/j.aprim.2017.11.003. Epub 2018 Feb 9. No abstract available. Spanish. PMID 29433757
- [Background] Miranda J, Underwood D, Kuepfer-Thomas M, Coulson D, Park AC, Butler SJ, Goldstein R, Brooks D, Everall AC, Guilcher SJT. Exploring transitions in care from pulmonary rehabilitation to home for persons with chronic obstructive pulmonary disease: A descriptive qualitative study. Health Expect. 2020 Apr;23(2):414-422. doi: 10.1111/hex.13012. Epub 2020 Jan 1. PMID 31893574
- [Background] Saavedra-Quiros V, Montero-Hernandez E, Menchen-Viso B, Santiago-Prieto E, Bermejo-Boixareu C, Hernan-Sanz J, Sanchez-Guerrero A, Campo Loarte J. [Medication reconciliation at admission and discharge. A consolidated experience]. Rev Calid Asist. 2016 Jun;31 Suppl 1:45-54. doi: 10.1016/j.cali.2016.02.002. Epub 2016 May 4. Spanish. PMID 27157795
- [Background] Gonzalez-Bueno J, Sevilla-Sanchez D, Puigoriol-Juvanteny E, Molist-Brunet N, Codina-Jane C, Espaulella-Panicot J. Improving medication adherence and effective prescribing through a patient-centered prescription model in patients with multimorbidity. Eur J Clin Pharmacol. 2022 Jan;78(1):127-137. doi: 10.1007/s00228-021-03207-9. Epub 2021 Aug 27. PMID 34448906
- [Background] Doos L, Bradley E, Rushton CA, Satchithananda D, Davies SJ, Kadam UT. Heart failure and chronic obstructive pulmonary disease multimorbidity at hospital discharge transition: a study of patient and carer experience. Health Expect. 2015 Dec;18(6):2401-12. doi: 10.1111/hex.12208. Epub 2014 May 16. PMID 24831061
- [Background] Hirschman KB, Shaid E, McCauley K, Pauly MV, Naylor MD. Continuity of Care: The Transitional Care Model. Online J Issues Nurs. 2015 Sep 30;20(3):1. PMID 26882510
- [Background] Arnar DO, Oddsson SJ, Gunnarsdottir T, Gudlaugsdottir GJ, Gudmundsson EF, Ketilsdottir A, Halldorsdottir H, Hrafnkelsdottir TJ, Hallsson H, Amundadottir ML, Thorgeirsson T. Improving outpatient care for heart failure through digital innovation: a feasibility study. Pilot Feasibility Stud. 2022 Nov 30;8(1):242. doi: 10.1186/s40814-022-01206-w. PMID 36451212
- [Background] Walker RC, Tong A, Howard K, Palmer SC. Patient expectations and experiences of remote monitoring for chronic diseases: Systematic review and thematic synthesis of qualitative studies. Int J Med Inform. 2019 Apr;124:78-85. doi: 10.1016/j.ijmedinf.2019.01.013. Epub 2019 Jan 29. PMID 30784430
- [Background] Coleman EA, Smith JD, Frank JC, Min SJ, Parry C, Kramer AM. Preparing patients and caregivers to participate in care delivered across settings: the Care Transitions Intervention. J Am Geriatr Soc. 2004 Nov;52(11):1817-25. doi: 10.1111/j.1532-5415.2004.52504.x. PMID 15507057
- [Background] Amblas-Novellas J, Martori JC, Molist Brunet N, Oller R, Gomez-Batiste X, Espaulella Panicot J. [Frail-VIG index: Design and evaluation of a new frailty index based on the Comprehensive Geriatric Assessment]. Rev Esp Geriatr Gerontol. 2017 May-Jun;52(3):119-127. doi: 10.1016/j.regg.2016.09.003. Epub 2016 Oct 28. Spanish. PMID 28029467
- [Background] Lavado A, Serra-Colomer J, Serra-Prat M, Burdoy E, Cabre M. Relationship of frailty status with health resource use and healthcare costs in the population aged 65 and over in Catalonia. Eur J Ageing. 2023 Jun 7;20(1):20. doi: 10.1007/s10433-023-00769-8. PMID 37280371
- [Background] Fernandez-Gasso L, Hernando-Arizaleta L, Palomar-Rodriguez JA, Abellan-Perez MV, Hernandez-Vicente A, Pascual-Figal DA. Population-based Study of First Hospitalizations for Heart Failure and the Interaction Between Readmissions and Survival. Rev Esp Cardiol (Engl Ed). 2019 Sep;72(9):740-748. doi: 10.1016/j.rec.2018.08.014. Epub 2018 Sep 24. English, Spanish. PMID 30262426
- [Background] Garcia Alcaraz F, Delicado Useros V, Alfaro Espin A, Lopez-Torres Hidalgo J. [The use of social healthcare resources and informal care characteristics care of immobilised homecare patients]. Aten Primaria. 2015 Apr;47(4):195-204. doi: 10.1016/j.aprim.2014.05.008. Epub 2014 Jul 11. Spanish. PMID 25027627
- [Background] Serra-Prat M, Moreno-Carmona MR, Fortuny A, Lavado A, Papiol M, Munoz L, Martinez-Cerda JF, Serra-Colomer J, Burdoy E, Cabre M. Frailty trends in Catalonia 2017-2021: An epidemiological study with 1.5 million people aged >/=65 years. Public Health. 2024 Dec;237:14-21. doi: 10.1016/j.puhe.2024.09.016. Epub 2024 Sep 23. PMID 39316851
- [Background] Laudicella M, Li Donni P, Smith PC. Hospital readmission rates: signal of failure or success? J Health Econ. 2013 Sep;32(5):909-21. doi: 10.1016/j.jhealeco.2013.06.004. Epub 2013 Jun 28. PMID 23938273
- [Background] S Alsulymani A, Ashram W, Alghamdi A, Hafiz HW, Ghunaim AM, Aljehani B, Aljabri A, Alzahrani G. Risk Factors for Readmission in Heart Failure Within 90 Days. Cureus. 2023 Dec 9;15(12):e50236. doi: 10.7759/cureus.50236. eCollection 2023 Dec. PMID 38084256
- [Background] Di Chiara C, Sartori G, Fantin A, Castaldo N, Crisafulli E. Reducing Hospital Readmissions in Chronic Obstructive Pulmonary Disease Patients: Current Treatments and Preventive Strategies. Medicina (Kaunas). 2025 Jan 9;61(1):97. doi: 10.3390/medicina61010097. PMID 39859079